CLINICAL TRIAL: NCT04016831
Title: Mapping Approaches to Prepare for Implementation Transfer (MAP-IT)
Acronym: MAP-IT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Jennifer Becan, Associate Research Scientist, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R21DA044261-02 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Mapping Approaches to Prepare for Implementation Transfer; Treatment Readiness and Induction Program

STUDY DESIGN:
Intervention Model Description: an implementation intervention to explore and address agency preparation needs in order to promote implementation success
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mapping Enhanced Counseling (MEC) only (Other): a motivational enhancement clinical intervention derived from cognitive-behavioral models that addresses problem recognition, treatment motivation, thoughtful and objective decision making, and therapeutic engagement
  Interventions: Behavioral: Mapping Enhanced Counseling (MEC)
- Mapping Approaches to Prepare for Implementation Transfer (Experimental): an implementation intervention to explore and address agency preparation needs in order to promote implementation success (includes MEC training)
  Interventions: Behavioral: Mapping Enhanced Counseling (MEC); Other: Mapping Approaches to Prepare for Implementation Transfer (MAP-IT)

INTERVENTIONS:
Behavioral: Mapping Enhanced Counseling (MEC) — a motivational enhancement clinical intervention derived from cognitive-behavioral models that addresses problem recognition, treatment motivation, thoughtful and objective decision making, and therapeutic engagement
Other: Mapping Approaches to Prepare for Implementation Transfer (MAP-IT) — an implementation intervention to explore and address agency preparation needs in order to promote implementation success
  Arms: Mapping Approaches to Prepare for Implementation Transfer

SUMMARY:
Despite demonstrated effectiveness, evidence based practices are not widely incorporated into existing residential and outpatient treatments. For implementation (and sustainment) of effective practices to be successful, it is critical that agencies be able to independently assess their own strengths and weaknesses and develop plans for organizational improvement. This application will extend scientific and field knowledge by providing a low-cost and sustainable alternative for improving agency preparedness for change.

DETAILED DESCRIPTION:
For implementation (and sustainment) of new interventions to be successful, it is critical that barriers are identified and addressed prior to change. It is challenging, however, for agencies to independently assess their own strengths and weaknesses and to develop plans for organizational improvement. Furthermore, the sheer number of strategies to promote implementation makes it difficult for agency leadership to decipher which are most appropriate for their own contexts and needs. This application proposes to develop and pilot test Mapping Approaches to Prepare for Implementation Transfer (MAP-IT), an organizational intervention that includes four key elements: (1) guidelines on forming an implementation workgroup to inform and promote implementation efforts, (2) instruction on mechanisms known to impact implementation, (3) tools and instruction for conducting an agency-driven diagnosis of potential implementation barriers, and (4) tools for developing an implementation blueprint to address identified barriers (including instruction on strategies for addressing potential barriers prior to implementation). The premise of this application is significant in that MAP-IT would provide a low-cost (agency-driven opportunity for deliberate implementation preparedness, without ongoing external coaching) and sustainable (skill development for multiple individuals within the organization that can be applied to future implementation efforts) alternative to promoting organizational adoption of new practices. The specific aims of the proposed research are as follows: Aim 1 - Synergistically integrate and adapt three established implementation intervention tools to promote deliberate agency implementation preparation - organizational assessment and feedback; taxonomy of implementation strategies; and visual-spatial decision making techniques - as combined into a comprehensive training and manualized bundle, MAP-IT. AIM 2 - Conduct a 2-arm cluster randomized efficacy trial of the MAP-IT intervention with 12 substance abuse treatment community-based residential and juvenile justice secure agencies serving adolescents (including those with opioid use disorders) randomized to either MAP-IT (EBP and MAP-IT trainings) or the non-intervention control condition (EBP training only). Successful completion of the aims is expected to (1) establish preliminary evidence for the efficacy of a low-cost, sustainable alternative for improving implementation preparation that agencies can use to support and expedite implementation transfer, (2) shift the current paradigm by encouraging researchers (designing uptake studies) and health care agencies (independently striving to implement new practices) to place greater emphasis on pre-implementation preparations for change, (3) provide an empirical examination of how exploration and preparation can support implementation, using established measurement platforms and theoretical frameworks, and (4) provide documentation of agency selection of implementation strategies for promoting change in real-world settings. Findings from the proposed R21 will inform intervention effectiveness testing and implementation strategy selection in a future R01 aimed at improving uptake of best practices within behavioral healthcare delivery services using a full-scale randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* clinical staff employed at adolescent substance use treatment agencies located in Texas with equal representation of community-based residential and secure justice agencies

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Preparation Intentions | Month 1, Month 2
  The proximal outcome (for hypothesis 1), preparation intentions (to address perceived implementation barriers through intentions to change organizational practices and use implementation strategies), is a continuous measure and will come from the TCU Workshop Evaluation Form (WEVAL).
Preparation Actions | Month 6
  The distal outcome (for hypothesis 2), preparation actions (to address perceived implementation barriers through changes in organizational practices and use of implementation strategies), is a continuous measure and will come from the TCU Workshop Assessment Follow-up Form (WAFU).
Organizational Climate | Baseline, Month 6
  The distal outcome (for hypothesis 3), organizational climate (change in mission, cohesion, autonomy, communication, stress, and proclivity to change), is 6 scale measures and will come from the TCU Survey of Organizational Functioning and Leadership (SOFL).
Staff Attributes | Baseline, Month 6
  The distal outcome (for hypothesis 3), staff attributes (change-oriented staff attributes including professional growth, efficacy, influence, and adaptability), is 4 scale measures and will come from the TCU Survey of Organizational Functioning and Leadership (SOFL).
Transformational Leadership | Baseline, Month 6
  The distal outcome (for hypothesis 3), transformational leadership (change in leader attributes including encourages innovation, inspirational motivation, develops others, and task delegation), is 4 scale measures and will come from the TCU Survey of Organizational Functioning and Leadership (SOFL).
Implementation Climate | Baseline, Month 6
  The distal outcome (for hypothesis 3), implementation readiness (pressure for change, organizational incentives and rewards, and leadership engagement in change process across time), is 3 scale measures and will come from the TCU Survey of Organizational Functioning and Leadership (SOFL).
Evidence Based Practice Attitude Scale (EBPAS) | Baseline, Month 6
  The distal outcome (for hypothesis 3), Evidence Based Practice Attitude Scale (EBPAS) is 4 scales to measure change in likelihood of adopting EBP given requirements to do so, intuitive appeal of EBP, openness to new practices, and perceived divergence of usual practice with research based/academically developed interventions.
EBP Implementation Adoption | Month 6
  The distal outcome (for hypothesis 4) measures adoption of the specified evidence-based practice (e.g., EBP sessions conducted).
EBP Penetration | Month 6
  The distal outcome (for hypothesis 4) measures penetration of the specified evidence-based practice (e.g., proportion of staff trained and using the EBP, proportion of clients receiving the EBP).
EBP Fidelity | Month 6
  The distal outcome (for hypothesis 4) measures implementation fidelity to the specified evidence-based practice (e.g., proportion of EBP sessions that adhered to core components).
Implementation Efficiency | Month 6
  The distal outcome (for hypothesis 5), implementation efficiency (e.g., time to prepare agency for implementation, train staff on the EBP, implement the EBP) is a continuous measure and will come from the Stages of Implementation Completion (SIC).

CONTACTS AND LOCATIONS:
Overall Officials: Jennfer R Becan, Ph.D., Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No